CLINICAL TRIAL: NCT05031013
Title: Trace Elements Concentration in Dialysis
Acronym: EMTDialyse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: laboratoire ILM - Université Lyon 1 CNRS, UMR 5306 UCBL (Unknown); MEXBrain 13 avenue Albert Einstein 69100 Villeurbanne (Unknown)
Responsible Party: Sponsor
Other Study IDs: 021ACR-EMTDialyse
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Dialysis
Keywords: dialysis; trace elements concentration; cadmium; lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — dialysat samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dialysis patients: Dialysis patients

SUMMARY:
In hemodialysis population the study team finds high concentrations of toxic trace elements (2 times higher than the general population for cadmium 4 to 13 times for lead). Several recent studies suggest a role of chronic exposure to cadmium in the loss of residual renal function, osteoporosis, graft failure, arteriosclerosis, as well as in excess cardiovascular mortality.

Moreover, in hemodialysis population, a deficit of certain essential trace elements (manganese, selenium, zinc) is observed. For example, in the population undergoing chronic hemodialysis, a zinc deficiency is found in 40 to 78% of cases. Zinc is a cofactor of more than 70 enzymes.

In this observational cohort, the study team seeks to understand the impact of HD and HDF on the serum concentrations of heavy metals and also oligometals, by studying their concentrations in the dialysate during dialysis sessions by inductive coupled plasma mass-spectrometry (ICP-MS).

DETAILED DESCRIPTION:
Primary objective: Evaluate the trace element concentration (heavy metals Cd and Pb and oligometals: Fe, Zn, Cu, Mn and also Se) in the dialysate before and during dialysis session. By studying the variation in concentration between the initial concentration of trace element in the dialysis fluid and the final concentration after membrane in the dialysate (waste pipe).

Method : Prospective study, in dialysis population, inclusion period will be from September 1, 2021 to January 31, 2022, in Ambroise Paré hospital, Paris, France. Duration of follow-up will be 1 day.

Dialysate samples will be taken in the venous injection site before connecting the patient, at 0 and 10 minutes after disinfection.

After connecting the patients, post-membrane dialysis sample (waste pipe) will be taken at 30, 60, 120 and 180minutes. Trace element dosage will be done by ICP-MS.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18;
* End-stage chronic renal failure in chronic dialysis;
* Duration of dialysis session ≥3h;
* Vascular approach: arteriovenous fistula;
* Affiliation to a social security scheme or entitled.

Exclusion Criteria:

* Opposition to participate to the study;
* Daily dialysis;
* Duration of dialysis session < 3h and > 8h;
* Vascular approach: venous catheter; Weekly dialysis session ≤3; Patient under french AME health system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Trace elements concentration | 5 months
  Trace elements concentration in the dialysate during dialysis sessions by inductive coupled plasma mass-spectrometry (ICP-MS).

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric Couturier, MD, Principal Investigator — Service néphrologie et dialyse, hôpital Ambroise Paré
Locations (1):
- Nephrology Department and Dialysis Unit, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonelli M, Wiebe N, Bello A, Field CJ, Gill JS, Hemmelgarn BR, Holmes DT, Jindal K, Klarenbach SW, Manns BJ, Thadhani R, Kinniburgh D; Alberta Kidney Disease Network. Concentrations of Trace Elements in Hemodialysis Patients: A Prospective Cohort Study. Am J Kidney Dis. 2017 Nov;70(5):696-704. doi: 10.1053/j.ajkd.2017.06.029. Epub 2017 Aug 31. PMID 28838766
- [Background] Prodanchuk M, Makarov O, Pisarev E, Sheiman B, Kulyzkiy M. Disturbances of trace element metabolism in ESRD patients receiving hemodialysis and hemodiafiltration. Cent European J Urol. 2014;66(4):472-6. doi: 10.5173/ceju.2013.04.art23. Epub 2014 Jan 27. PMID 24757548
- [Background] Orr SE, Bridges CC. Chronic Kidney Disease and Exposure to Nephrotoxic Metals. Int J Mol Sci. 2017 May 12;18(5):1039. doi: 10.3390/ijms18051039. PMID 28498320
- [Background] Messner B, Knoflach M, Seubert A, Ritsch A, Pfaller K, Henderson B, Shen YH, Zeller I, Willeit J, Laufer G, Wick G, Kiechl S, Bernhard D. Cadmium is a novel and independent risk factor for early atherosclerosis mechanisms and in vivo relevance. Arterioscler Thromb Vasc Biol. 2009 Sep;29(9):1392-8. doi: 10.1161/ATVBAHA.109.190082. Epub 2009 Jun 25. PMID 19556524
- [Background] Lee CC, Weng CH, Huang WH, Yen TH, Lin JL, Lin-Tan DT, Chen KH, Hsu CW. Association Between Blood Cadmium Levels and Mortality in Peritoneal Dialysis. Medicine (Baltimore). 2016 May;95(19):e3717. doi: 10.1097/MD.0000000000003717. PMID 27175714
- [Background] Sotomayor CG, Groothof D, Vodegel JJ, Eisenga MF, Knobbe TJ, IJmker J, Lammerts RGM, de Borst MH, Berger SP, Nolte IM, Rodrigo R, Slart RHJA, Navis GJ, Touw DJ, Bakker SJL. Plasma cadmium is associated with increased risk of long-term kidney graft failure. Kidney Int. 2021 May;99(5):1213-1224. doi: 10.1016/j.kint.2020.08.027. Epub 2020 Sep 14. PMID 32941876
- [Background] Larsson SC, Wolk A. Urinary cadmium and mortality from all causes, cancer and cardiovascular disease in the general population: systematic review and meta-analysis of cohort studies. Int J Epidemiol. 2016 Jun;45(3):782-91. doi: 10.1093/ije/dyv086. Epub 2015 May 20. PMID 25997435
- [Background] Satarug S, C Gobe G, A Vesey D, Phelps KR. Cadmium and Lead Exposure, Nephrotoxicity, and Mortality. Toxics. 2020 Oct 13;8(4):86. doi: 10.3390/toxics8040086. PMID 33066165
- [Background] Roozbeh J, Sharifian M, Sagheb MM, Shabani S, Hamidian Jahromi A, Afshariani R, Pakfetrat M, Salehi O. Comment on: does zinc supplementation affect inflammatory markers in hemodialysis patients? Ren Fail. 2011;33(4):466-7. doi: 10.3109/0886022X.2011.568144. No abstract available. PMID 21529280